CLINICAL TRIAL: NCT06776627
Title: Effectiveness of an Adapted Physical Activity Program on Improving the Health-related Quality of Life of Women With Endometriosis in Martinique
Acronym: APAENDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: ARGOS (Association pour la Recherche en Gynécologie Obstétrique et Stérilité) (Unknown); SAPHYR Martinique (Association Santé par l'activité physique régulière) (Unknown); ECM Rénovbat (Unknown); Agence Régionale de Santé de la Martinique (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24_RIPH2-03; 2024-A01875-42 (Other: ID-RCB)
Record Dates: First submitted 2024-11-27; First posted 2025-01-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis
Keywords: Endometriosis; Adapted physical activity; Quality of life
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine care (No Intervention): 31 patients: Routine consultation including:
  * clinical examination
  * pain scale
  * ECG
  * vital signs
  * fat and muscle mass
  * medical history
  * biological assessment
  * quality of life questionnaire (EHP-30)
  * sedentary lifestyle and physical activity test
  * sleep scale (PSQI)
- Routine care + adapted physical activity (APA) (Experimental): Patients randomized to the APA group will be prescribed, at the end of the routine consultation, 12 weeks of adapted physical activity sessions, to be carried out outdoors, and coordinated by a qualified professional from the STAPS sector (Master's degree in Science and Technology of Physical and Sporting Activities). The latter will provide patients with an adapted program determined following a personalized physical condition assessment: aerobic capacity, strength, endurance, flexibility, balance and proprioception tests.
  Interventions: Other: Adapted physical activity (APA)

INTERVENTIONS:
Other: Adapted physical activity (APA) — Adapted program: aerobic capacity, strength, endurance, flexibility, balance and proprioception tests. APA sessions take place over 12 weeks. There will be 2 to 3 sessions per week. Course of a session: - Warm-up: 10-15min: cycling or walking. - Moderate-intensity endurance activity: cycling, walking or swimming: 10min, the duration will be increased gradually up to a minimum of 30min at the end of the program. - Muscle strengthening: with polyarticular or monoarticular exercises targeting the upper limbs or lower limbs in alternation and sheathing. At the beginning: 8 exercises per session and 8 repetitions, 1 time per week. Objective will be to increase the number of repetitions and then integrate other exercises to reach 10 exercises with 12 repetitions, 2 times per week. - Stretching and balance: learning to stretch the muscle groups worked and then working on proprioception (bipodal, monopodal station, then double task). - Quiet time: relaxation through breathing 5 min.
  Arms: Routine care + adapted physical activity (APA)

SUMMARY:
There is no specific treatment for endometriosis, because the pathophysiology is poorly understood.

Adapted physical activity (APA) is recognized as a beneficial supportive care for patients suffering from chronic pathology. Adapted physical activity can play a role in managing endometriosis symptoms. Studies have shown that regular physical exercise can help reduce pain, improve quality of life and alleviate symptoms related to chronic diseases.

However, it is known that few women with endometriosis have regular physical activity because of pain, chronic fatigue that lead to activity limitation or even disability.

This study provides an opportunity to evaluate the impact of regular APA practice on improving the quality of life and symptoms of women with endometriosis in Martinique.

Based on this, APA could be included in the endometriosis care pathway in Martinique.

DETAILED DESCRIPTION:
The investigators' hypothesis is that APA improves the overall quality of life of women with endometriosis and also has a positive impact on pain, functional abilities and sleep. The effectiveness of the proposed adapted physical activity program also improves the psycho-social and professional impact of the disease in the daily lives of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman of childbearing age,
* Clinico-radiological or clinico-histological diagnosis of endometriosis: laparoscopy with biopsy or MRI,
* History of endometriosis symptoms before diagnosis,
* Walking without technical assistance,
* Able to read and write,
* Patient wishing to improve her health by optimizing her lifestyle,
* Patient affiliated or beneficiary of a social security scheme,
* Patient having given free, informed and written consent.

Exclusion Criteria:

* Acute or terminal illness,
* Recent fracture of the upper or lower limbs (< 3 months),
* Other chronic unstable or orthopedic illness that could interfere with the ability to participate in a physical activity program,
* Resting ECG at inclusion outside the normal range,
* Patients who practice moderate to intense physical activity for more than 150 minutes per week,
* Absolute contraindication to physical activity linked to severe co-morbidities,
* Patient placed under legal protection, guardianship or curatorship,
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness at 12 weeks of an adapted physical activity program on the health-related quality of life of patients with endometriosis. | 12 weeks
  The level of health-related quality of life will be measured using the EHP-30 (Endometriosis Health Profile) questionnaire.
  The minimum value is 0, and the maximum value is 100. Higher score mean a worse outcome.

SECONDARY OUTCOMES:
To evaluate the effectiveness at 9 weeks of an adapted physical activity program in patients with endometriosis on health-related quality of life. | 12 weeks
  The level of health-related quality of life will be measured using the EHP-30 (Endometriosis Health Profile) questionnaire. The minimum value is 0, and the maximum value is 100. Higher score mean a worse outcome.
To evaluate the effectiveness at 9 and 12 weeks of an adapted physical activity program in patients with endometriosis on improvement of pain | 12 weeks
  Pain will be assessed by the Visual Analogue Scale. The minimum value is 0 cm, and the maximum value is 10 cm. Higher score mean a worse outcome.
To evaluate the effectiveness at 9 and 12 weeks of an adapted physical activity program in patients with endometriosis on improvement of functional capacities of physical condition, and activity level | 12 weeks
  Assessed by the Ricci and Gagnon questionnaire. The minimum value is 9, and the maximum value is 45. Higher score mean a better outcome.
To evaluate the effectiveness at 9 and 12 weeks of an adapted physical activity program in patients with endometriosis on improving sleep quality | 12 weeks
  Sleep quality with the questionnaire: PSQI (Pittsburgh Sleep Quality Index). The minimum value is 0, and the maximum value is 21. Higher score mean a worse outcome.
To evaluate the effectiveness at 9 and 12 weeks of an adapted physical activity program in patients with endometriosis on improving the professional, psychosocial impact of the disease in the daily lives of patients | 12 weeks
  The psycho-socio-family and professional impact by using the part 2 of the EHP-30 (Endometriosis Health Profile) (section A and B).
To evaluate the effectiveness at 9 and 12 weeks of an adapted physical activity program in patients with endometriosis on improvement of grip muscle strength, flexibility, walking perimeter, and physical profile | 12 weeks
  Functional capacities of physical condition: measurement of blood pressure.
To evaluate the effectiveness at 9 and 12 weeks of an adapted physical activity program in patients with endometriosis on improvement of grip muscle strength, flexibility, walking perimeter, and physical profile | 12 weeks
  Functional capacities of physical condition: measurement of heart rate.
To evaluate the effectiveness at 9 and 12 weeks of an adapted physical activity program in patients with endometriosis on improvement of grip muscle strength, flexibility, walking perimeter, and physical profile | 12 weeks
  Functional capacities of physical condition: grip muscle strength (hand grip).
To evaluate the effectiveness at 9 and 12 weeks of an adapted physical activity program in patients with endometriosis on improvement of grip muscle strength, flexibility, walking perimeter, and physical profile | 12 weeks
  Functional capacities of physical condition: measurement of flexibility: with finger/ground distance.
To evaluate the effectiveness at 9 and 12 weeks of an adapted physical activity program in patients with endometriosis on improvement of grip muscle strength, flexibility, walking perimeter, and physical profile | 12 weeks
  Functional capacities of physical condition: measurement of walking capacity with the 6-minute walk test.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Center of Martinique, Fort-de-France, Martinique, France

IPD SHARING:
Plan to Share IPD: No